CLINICAL TRIAL: NCT06907667
Title: Study of the Impact of Time of Vaccination on Response to Influenza Vaccine in Patients With Chronic Renal Failure - CHRONOVAX 2
Brief Title: Study of the Impact of Time of Vaccination on Response to Influenza Vaccine in Patients With Chronic Renal Failure
Acronym: CHRONOVAX2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-API-01
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Vaccination; Infection
Keywords: Influenza; chronic renal insufficiency; Vaccination
MeSH Terms: conditions — Infections; Influenza, Human; Renal Insufficiency, Chronic | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning injection (Active Comparator): VAXIGRIPTETRA influenza vaccine injection between 07:00 am and 11:00 am.
  Interventions: Other: Vaccine injection
- Evening injection (Active Comparator): VAXIGRIPTETRA influenza vaccine injection between 05:00 pm and 09:00 pm.
  Interventions: Other: Vaccine injection

INTERVENTIONS:
Other: Vaccine injection — Injection of the vaccine in chronic renal insufficiency patients.
  Other Names: VAXIGRIPTETRA - quadrivalent inactivated influenza vaccine.

SUMMARY:
Immune response to influenza vaccine in patients with chronic renal insufficiency.

DETAILED DESCRIPTION:
Seasonal influenza vaccination is recommended for patients with chronic renal insufficiency, as influenza is responsible for significant morbidity and mortality in this immunocompromised population. However, the immune response to this vaccination is limited in this population.

There are currently no recommendations concerning the timing of influenza vaccine in the general population or in immunocompromised patients.

In this context, recent studies have shown that the time of vaccination can have an impact on vaccine efficacy. This is the case for BCG, influenza and COVID vaccinations.

On this basis, our main hypothesis is that the administration of influenza vaccine to patients with chronic kidney failure is more effective in the morning than in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patient at stage 4 or 5 (i.e. estimated GFR < 30mL/min/1.73m2); or Dialysis patient; or renal transplant patient regardless of GFR;
* Age ≥ 18 years;
* Indication for influenza vaccination;
* Express free and informed consent.

Exclusion Criteria:

* Known hypersensitivity to influenza vaccine or egg proteins;
* Previous influenza vaccination for the current season;
* Current infection;
* Current acute illness;
* Treatments with a major impact on vaccine response:
* Treatment of rejection within the previous 3 months;
* Renal transplantation with induction performed within the previous 6 months;
* Immunosuppressive treatment including CTLA4 agonist, complement inhibitor, anti-CD20;
* Treatments that may distort the serological response: Polyvalent immunoglobulin infusion within the preceding 3 months;
* Vulnerable persons (minors, adults under guardianship or trusteeship, persons deprived of their liberty, persons unable to speak French);
* Subjects not affiliated to Social Security.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Antibody titers (seroconversion) at 4 weeks after injection of inactivated influenza vaccine in each arm. | 7 months
  Seroconversion will be defined as an increase in antibody titer of at least 4-fold (≥4) over pre-vaccination titer AND an antibody titer ≥ 1:40 (seroprotection) four weeks post-vaccination, for at least one of the three vaccine antigens.

SECONDARY OUTCOMES:
Number of seasonal influenza virus infections in each arm at 4 weeks | 7 months
  Comparing the number of seasonal influenza virus infections in each arm between a group of patients vaccinated in the morning and a group vaccinated in the evening at 4 weeks.
  The occurrence of influenza, as confirmed by a PCR test, will be noted in the follow-up consultation.
Number of seasonal influenza virus infections in patients with chronic renal insufficiency at 6 months | 12 months
  Comparing the number of seasonal influenza virus infections in patients with chronic renal failure between a group of patients vaccinated in the morning and a group vaccinated in the evening in the 6 months following vaccination.
  The occurrence of influenza, as confirmed by a PCR test, will be noted in the follow-up consultation.
Antibody titers reacting in each arm | 7 months
  In patients with chronic renal failure, compare the evolution of antibody titres reacting with vaccine antigens 4 weeks after influenza vaccination between a group of patients vaccinated in the morning and a group of patients vaccinated in the evening.
  The titer of antibodies reacting with vaccine antigens is measured by ELISA ;
Number of anti-vaccine antibodies inhibiting hemmagglutination | 7 months
  4 weeks after influenza vaccine injection, compare hemmagglutination-inhibiting anti-vaccine antibody titer in CKD patients vaccinated in the morning and evening.
  The titer of hemagglutination-inhibiting anti-vaccine antibodies will be determined by hemagglutination inhibition test
Number of neutralizing anti-vaccine antibodies | 7 months
  To compare, 4 weeks after influenza vaccine injection, the titer of neutralizing antivaccine antibodies in CKD patients vaccinated in the morning and evening.
  The titer of neutralizing anti-vaccine antibodies will be determined by a pseudo-neutralization test.

CONTACTS AND LOCATIONS:
Overall Officials: GOSSET Clément, MD, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice - Hôpital Pasteur 2, Nice, Alpes-Maritimes, France